CLINICAL TRIAL: NCT00740610
Title: A Phase 2, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Activity of GS 9450 in Adults With Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Safety, Tolerability, Pharmacokinetics and Activity of GS-9450 in Adults With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-228-0101
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): 22 subjects to receive 1 mg GS-9450 for 4 weeks
  Interventions: Drug: GS-9450
- Cohort 2 (Experimental): 22 subjects to receive 5 mg GS-9450 for 4 weeks
  Interventions: Drug: GS-9450
- Cohort 3 (Experimental): 22 subjects to receive 10 mg GS-9450 for 4 weeks
  Interventions: Drug: GS-9450
- Cohort 4 (Experimental): 22 subjects to receive 40 mg GS-9450 for 4 weeks
  Interventions: Drug: GS-9450
- Cohort 5 (Placebo Comparator): 22 subjects to receive placebo to match GS-9450 for 4 weeks
  Interventions: Drug: GS-9450 Placebo

INTERVENTIONS:
Drug: GS-9450 — GS-9450 capsules at a dose of 1, 5, 10, and 40 mg administered orally once daily
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Drug: GS-9450 Placebo — Placebo to match GS-9450 administered orally once daily
  Arms: Cohort 5

SUMMARY:
The overall purpose of this study is to examine the safety, tolerability, pharmacokinetics (how the body processes a drug), and activity of GS-9450 in preventing liver damage due to scarring, or fibrosis, caused by Non-Alcoholic Steatohepatitis (also known as NASH).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, parallel group, placebo controlled, multicenter study investigating the safety, tolerability, pharmacokinetics and activity of multiple oral doses of GS 9450 in adults with NASH. Approximately 110 subjects 18 75 years of age with elevated ALT (> 60 U/L at screening), fatty liver on screening ultrasound, and biopsy-proven NASH will be randomized (1:1:1:1:1) to one of five parallel treatment groups (22 subjects per treatment group) as follows:

GS-9450 1mg by mouth (PO) once daily, GS-9450 5 mg PO once daily, GS-9450 10 mg PO once daily, GS-9450 40 mg PO once daily, or Matching placebo PO once daily Qualifying subjects will be stratified by the presence/absence of type 2 diabetes (i.e., on/off oral diabetic medication at entry) and by geographic region (US and France). Following randomization, subjects will return within five business days later for a baseline visit, at which time they will be dispensed study medication and enter a 4-week treatment phase. Upon completion of the treatment phase, subjects will enter a 4 week off-treatment follow-up period. Each subject's participation in the study will last up to approximately 12 weeks (inclusive of screening, treatment phase, and off-treatment follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* ALT > 60 U/L
* fatty liver on screening ultrasound
* and biopsy-confirmed NASH
* platelet count >/= 75,000/mm3 and adequate hematologic function (absolute neutrophil count >/= 1,500/mm3, hemoglobin >/= 11.0 g/dL)
* calculated creatinine clearance >/= 70 mL/min
* non-insulin dependent diabetes for < 10 years is allowed if stably managed for at least 6 months prior to screening
* stable weight (no weight loss > 4%) for 8 weeks prior to screening and should maintain consistent diet, food intake, and physical exercise during the study
* must have been on stable therapy for at least 3 months prior to screening if receiving 3-hydroxy-3-methylglutaryl-coenzyme (HMG-CoA) reductase inhibitors, niacin, fibrates, vitamin E or angiotensin receptor blockers
* must have been on a stable treatment regimen for at least 3 months prior to screening if receiving other drugs possibly associated with hepatic adverse events (e.g., isoniazid, itraconazole, ketoconazole, rifabutin, rifampin, and other agents with significant hepatotoxic potential)

Exclusion Criteria:

* Insulin dependent diabetes mellitus, treatment with sulfonylureas (may be allowed pending results from a drug-drug interaction study), subjects receiving glitazones at screening or within 6 months of screening, presence of diabetic peripheral neuropathy or gastroparesis
* A > 4% decrease in weight within 8 weeks of screening
* cirrhosis or decompensated liver disease (defined as conjugated bilirubin > 1.5 x the upper limit of the normal range (ULN), prothrombin time > 1.5 x ULN, serum albumin < 3.0 g/dL, or prior history of clinical hepatic decompensation
* presence of other form of liver disease other than NASH
* history of excess alcohol ingestion, averaging > 3 drinks/day in the previous 2 years; or current alcohol intake averaging > 2 drinks/day for females and > 3 drinks per day for males; history of or current binge drinking
* serological evidence of co-infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV
* evidence of hepatocellular carcinoma (i.e., α-fetoprotein > 50 ng/mL)
* history of ingesting drugs possibly associated with hepatic steatosis within the past year
* history of total parenteral nutrition within the past 6 months
* prior history of gastroplasty, jejunoileal, or jejunocolonic bypass surgery
* history of ingesting drugs within the past 3 months that may improve NASH and associated fibrosis
* significant gastrointestinal disease that would interfere with absorption of oral medications; inflammatory bowel disease
* major surgery within the past year
* clinically significant abnormalities on ECG or other ECG findings that the investigator considers a safety risk
* significant systemic or major illnesses other than liver disease that, in the opinion of the investigator, would preclude treatment and adequate follow up
* prior or current malignancy involving any organ system and skin cancer (previously excised basal cell carcinoma allowed)
* acute ongoing infection, or symptoms of infection
* pregnant or breastfeeding females
* acute substance abuse within the past year.
* history of ingesting anti-TNFα drugs or immunomodulators within the past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced Adverse Events (AEs) and Graded Laboratory Abnormalities | Baseline to Post-treatment Week 24

SECONDARY OUTCOMES:
Pharmacokinetics of GS-9450 and its metabolites | Weeks 2 and 4
  Pharmacokinetics (Cmax, Tmax, Cmin, λz, t1/2, AUCtau, Vdss/F, and CL/F) measured by plasma sampling
Change from baseline in alanine aminotransferase (ALT) | Baseline to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Mondou, MD, Study Director — Gilead Sciences
Locations (33):
- United States (31):
  - Tucson, Arizona
  - Fresno, California
  - Fullerton, California
  - San Diego, California
  - San Mateo, California
  - Lakewood, Colorado
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Troy, Michigan
  - New York, New York
  - Plainview, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Clevleand, Ohio
  - Providence, Rhode Island
  - Dallas, Texas
  - Galveston, Texas
  - Irving, Texas
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Richmond, Virginia
- France (2):
  - Paris
  - Vandœuvre-lès-Nancy